CLINICAL TRIAL: NCT05032690
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, 3-PERIOD, 4-SEQUENCE, CROSSOVER, SINGLE-DOSE STUDY TO COMPARE THE BIOAVAILABILITY OF ORALLY ADMINISTERED BOSUTINIB CAPSULES AND TO ESTIMATE THE EFFECT OF FOOD ON BOSUTINIB CAPSULE
Brief Title: Evaluation of the Relative Bioavailability of Bosutinib Capsules Under Fed Condition and Estimation of Food Effect on Orally Administered Bosutinib Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B1871062; 2021-004911-24 (EudraCT Number)
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-05

CONDITIONS: Healthy Participants
Keywords: Bioavailability; Food Effect; Bosutinib; Maximum Observed Plasma Concentration (Cmax); Area Under the Curve (AUC)
MeSH Terms: interventions — bosutinib

STUDY DESIGN:
Intervention Model Description: A Phase 1, open-label, randomized, single dose, 3-period, 4 sequence, crossover study in healthy participants
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment B: Bosutinib four 25 mg capsule after meal (Experimental): Bosutinib four 25 mg capsule taken after a high-fat and high-calorie breakfast for comparison 1
  Interventions: Drug: Bosutinib capsule
- Treatment A: Bosutinib 100 mg capsule after meal (active comparator) (Active Comparator): Bosutinib 100 mg capsule taken after a high-fat and high-calorie breakfast for comparison 1
  Interventions: Drug: Bosutinib capsule
- Treatment A: Bosutinib 100 mg capsule after meal (experimental) (Experimental): Bosutinib 100 mg capsule taken after a high-fat and high-calorie breakfast for comparison 2
  Interventions: Drug: Bosutinib capsule
- Treatment C: Bosutinib 100 mg capsule after fasting (Active Comparator): Bosutinib 100 mg capsule taken after an overnight fast of at least 10 hours for comparison 2
  Interventions: Drug: Bosutinib

INTERVENTIONS:
Drug: Bosutinib capsule — Bosutinib four 25 mg capsule taken after a high-fat and high calorie breakfast
  Arms: Treatment B: Bosutinib four 25 mg capsule after meal
Drug: Bosutinib capsule — Bosutinib 100 mg capsule taken after a high-fat and high calorie breakfast
  Arms: Treatment A: Bosutinib 100 mg capsule after meal (active comparator)
Drug: Bosutinib — Bosutinib 100 mg capsule taken after an overnight fast of at least 10 hours
  Arms: Treatment C: Bosutinib 100 mg capsule after fasting
Drug: Bosutinib capsule — Bosutinib 100 mg capsule taken after a high-fat and high-calorie breakfast
  Arms: Treatment A: Bosutinib 100 mg capsule after meal (experimental)

SUMMARY:
This study is intended to estimate the bioavailability of a single 100 mg bosutinib capsules relative to four 25 mg capsules under fed condition in adult healthy participants and to estimate the effect of a high-fat, high-calorie meal on the bioavailability of a single 100 mg capsule of bosutinib relative to fasted condition in adults healthy participants. The comparisons will be performed using the pharmacokinetic parameters that define the rate and extend of absorption (Cmax, AUC). Statistical analyses will be performed after the administration of a single 100 mg dose under fed condition as the Reference treatment and the four 25 mg capsules as the Test treatment for the first comparison, and after administration of a single 100 mg dose under fasted condition as the Reference treatment and the 100 mg capsule under fed condition as the Test treatment for the second comparison.

ELIGIBILITY:
Inclusion Criteria:

* Female participants of non-childbearing potential and/or male participants must be 18 to 55 years of age, inclusive, at the time of signing the informed consent document (ICD)
* participants who are overtly healthy as determined by medical evaluation including a detailed medical history, complete physical examination, vital signs which include BP and pulse rate measurement, clinical laboratory tests, and electrocardiogram (ECG).
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological, or allergic disease.
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg,hepatitis B surface antigen (HBcAb) or hepatitis C antibody (HCVAb).
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study-specific laboratory and confirmed by a single repeat test, if deemed necessary:

  * estimated glomerular filtration rate (eGFR) (Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]) <90 mL/min/1.73 m2;
  * aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level >upper limit of normal (ULN);
  * Serum (total and direct) bilirubin level > ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is <= ULN;
  * Amylase and lipase level > ULN.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1871062

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 32 participants were assigned to the study intervention, of whom 26 participants received all the randomized treatment by sequence and 25 participants completed the study.
Groups:
- Treatment A -> Treatment B -> Treatment C: Treatment A: 1 × 100 mg bosutinib capsule under fed condition. Treatment B: 4 × 25 mg bosutinib capsules under fed condition. Treatment C: 1 × 100 mg bosutinib capsule under fasted condition. The participant took Treatment A in Period 1, followed with at least 14-days washout between successive bosutinib doses, and then Treatment B in Period 2, followed with another at least 14-days washout between successive bosutinib doses, and then Treatment C in Period 3.
- Treatment B -> Treatment A -> Treatment C: Treatment A: 1 × 100 mg bosutinib capsule under fed condition. Treatment B: 4 × 25 mg bosutinib capsules under fed condition. Treatment C: 1 × 100 mg bosutinib capsule under fasted condition. The participant took Treatment B in Period 1, followed with at least 14-days washout between successive bosutinib doses, and then Treatment A in Period 2, followed with another at least 14-days washout between successive bosutinib doses, and then Treatment C in Period 3.
- Treatment A ->Treatment B: Treatment A: 1 × 100 mg bosutinib capsule under fed condition. Treatment B: 4 × 25 mg bosutinib capsules under fed condition.The participant took Treatment A in Period 1, followed with at least 14-days washout between successive bosutinib doses, and then Treatment B in Period 2.
- Treatment B->Treatment A: Treatment A: 1 × 100 mg bosutinib capsule under fed condition. Treatment B: 4 × 25 mg bosutinib capsules under fed condition. The participant took Treatment B in Period 1, followed with at least 14-days washout between successive bosutinib doses, and then Treatment A in Period 2.
Period: Period 1
Arm/Group | Treatment A -> Treatment B -> Treatment C | Treatment B -> Treatment A -> Treatment C | Treatment A ->Treatment B | Treatment B->Treatment A
Started | 8 | 10 | 7 | 7
Completed | 7 | 8 | 7 | 7
Not Completed | 1 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — No longer meets eligibility criteria | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | Treatment A -> Treatment B -> Treatment C | Treatment B -> Treatment A -> Treatment C | Treatment A ->Treatment B | Treatment B->Treatment A
Started | 7 | 8 | 7 | 7
Completed | 6 | 6 | 7 | 7
Not Completed | 1 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — No longer meets eligibility criteria | 0 | 1 | 0 | 0
Period: Period 3
Arm/Group | Treatment A -> Treatment B -> Treatment C | Treatment B -> Treatment A -> Treatment C | Treatment A ->Treatment B | Treatment B->Treatment A
Started | 6 | 6 | 0 | 0
Completed | 6 | 5 | 0 | 0
Not Completed | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A -> Treatment B -> Treatment C | Treatment B -> Treatment A -> Treatment C | Treatment A ->Treatment B | Treatment B->Treatment A | Total
Number analyzed (Participants) | 8 | 10 | 7 | 7 | 32
Age, Continuous [Median (Full Range); unit: years] | 35.5 [19 to 54] | 38.0 [23 to 53] | 42.0 [23 to 49] | 42.0 [22 to 47] | 39.5 [19 to 54]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8 | 10 | 7 | 7 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 8 | 10 | 6 | 6 | 30
  Hispanic or Latino | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUCinf) for Bosutinib
Description: AUCinf was calculated as [AUClast+(Clast*/kel)], where AUClast is the area under the plasma concentration-time profile from time 0 to the time of the Clast, Clast is the last quantifiable concentration, Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis, and kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. The geometric coefficient of variation was reported as percentage
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: The pharmacokinetic (PK) parameter analysis population is defined as all subjects randomized and treated who have at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Treatment A: Bosutinib 1*100 mg Capsule Fed: Following an overnight fast of at least 10 hours and after the collection of predose bosutinib PK sample on Day 1, participants will receive a high-fat, high-calorie breakfast approximately 30 minutes prior to dosing which should be completed within approximately 20 minutes. The participants received 100 mg capsule of bosutinib at approximately 0800 hours (±2 hours), approximately 10 minutes after the completion of the breakfast.
- Treatment B: Bosutinib 4*25 mg Capsule Fed: Following an overnight fast of at least 10 hours and after the collection of predose bosutinib PK sample on Day 1, participants received a high-fat, high-calorie breakfast approximately 30 minutes prior to dosing which should be completed within approximately 20 minutes. The participants will then receive 4*25 mg capsule of bosutinib at approximately 0800 hours (±2 hours), approximately 10 minutes after the completion of the breakfast.
- Treatment C: Bosutinib 1*100 mg Capsule Fasted: Following an overnight fast of at least 10 hours and after the collection of predose bosutinib PK sample on Day 1, participants received 100 mg capsule of bosutinib at approximately 0800 hours (±2 hours).
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
Number analyzed (Participants) | 21 | 20 | 4
nanogram*hour per milliliter (ng*hr/mL) | 591.3 (32) | 591.7 (39) | 479.4 (30)
Statistical Analysis 1: Comparison: Treatment A: Bosutinib 1*100 mg Capsule Fed vs Treatment B: Bosutinib 4*25 mg Capsule Fed; For comparison of Bosutinib 4*25 mg Capsule Fed vs. Bosutinib 1*100 mg Capsule Fed, the model is a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The reference treatment of Bosutinib 4*25 mg Capsule Fed is Bosutinib 1*100 mg Capsule Fed; Test type: Equivalence — The adjusted mean differences and 90% CIs for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% CIs for the ratios. The ratio of adjusted geometric means and 90% confidence interval were expressed as percentages; Mixed Models Analysis; ratio of adjusted geometric means = 99.17, 90% CI 2-sided [93.72 to 104.93]
Statistical Analysis 2: Comparison: Treatment A: Bosutinib 1*100 mg Capsule Fed vs Treatment C: Bosutinib 1*100 mg Capsule Fasted; For comparison of Bosutinib 1*100 mg Capsule Fed vs. Bosutinib 1*100 mg Capsule Fasted, the model is a mixed effect model with sequence and treatment as fixed effects and participant within sequence as a random effect. The reference treatment of Bosutinib 1*100 mg Capsule Fed is Bosutinib 1*100 mg Capsule Fasted; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; ratio of adjusted geometric means = 135.90, 90% CI 2-sided [109.28 to 169.01]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) for Bosutinib
Description: Cmax was the maximum observed plasma concentration. The geometric coefficient of variation was reported as percentage.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: The PK parameter analysis population is defined as all subjects randomized and treated who have at least 1 of the PK parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Treatment A: Bosutinib 1*100 mg Capsule Fed: Following an overnight fast of at least 10 hours and after the collection of predose bosutinib PK sample on Day 1, participants will receive a high-fat, high-calorie breakfast approximately 30 minutes prior to dosing which should be completed within approximately 20 minutes. The participants will then receive 100mg capsule of bosutinib at approximately 0800 hours (±2 hours), approximately 10 minutes after the completion of the breakfast.
- Treatment B: Bosutinib 4*25 mg Capsule Fed: Following an overnight fast of at least 10 hours and after the collection of predose bosutinib PK sample on Day 1, participants will receive a high-fat, high-calorie breakfast approximately 30 minutes prior to dosing which should be completed within approximately 20 minutes. The participants will then receive 4*25 mg capsule of bosutinib at approximately 0800 hours (±2 hours), approximately 10 minutes after the completion of the breakfast.
- Treatment C: Bosutinib 1*100 mg Capsule Fasted: Following an overnight fast of at least 10 hours and after the collection of predose bosutinib PK sample on Day 1, participants will receive 100 mg capsule of bosutinib at approximately 0800 hours (±2 hours).
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
Number analyzed (Participants) | 30 | 31 | 12
nanogram per milliliter (ng/mL) | 17.80 (40) | 16.68 (38) | 10.75 (58)
Statistical Analysis 1: Comparison: Treatment A: Bosutinib 1*100 mg Capsule Fed vs Treatment B: Bosutinib 4*25 mg Capsule Fed; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; ratio of adjusted geometric means = 93.77, 90% CI 2-sided [90.08 to 97.61]
Statistical Analysis 2: Comparison: Treatment A: Bosutinib 1*100 mg Capsule Fed vs Treatment C: Bosutinib 1*100 mg Capsule Fasted; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; ratio of adjusted geometric means = 162.54, 90% CI 2-sided [130.25 to 202.84]

3. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) for Bosutinib
Description: AUClast was the area under the concentration-time curve from time 0 to the time of the last quantifiable concentration.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
Number analyzed (Participants) | 30 | 31 | 12
nanogram*hour per milliliter (ng*hr/mL) | 455.6 (40) | 446.4 (45) | 301.6 (52)
Statistical Analysis 1: Comparison: Treatment A: Bosutinib 1*100 mg Capsule Fed vs Treatment B: Bosutinib 4*25 mg Capsule Fed; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; ratio of adjusted geometric means = 98.21, 90% CI 2-sided [93.83 to 102.80]
Statistical Analysis 2: Comparison: Treatment A: Bosutinib 1*100 mg Capsule Fed vs Treatment C: Bosutinib 1*100 mg Capsule Fasted; [analysis description as in outcome 1, analysis 2]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; ratio of adjusted geometric means = 146.70, 90% CI 2-sided [117.88 to 182.58]

4. Secondary Outcome: Time for Cmax (Tmax) of Bosutinib
Description: Tmax was the time to reach maximum observed plasma concentration and was observed directly from data as time of the first occurrence.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
Number analyzed (Participants) | 30 | 31 | 12
hour | 6.00 [4.00 to 12.00] | 6.00 [3.00 to 8.00] | 6.00 [3.00 to 8.02]

5. Secondary Outcome: Apparent Clearance After Oral Dose (CL/F) of Bosutinib
Description: CL/F was the apparent clearance after oral dose and was determined as dose/AUCinf. The geometric coefficient of variation was reported as percentage.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
Number analyzed (Participants) | 21 | 20 | 4
liter/hour | 169.3 (32) | 169.0 (39) | 208.5 (30)

6. Secondary Outcome: Apparent Volume of Distribution After Oral Dose (Vz/F) of Bosutinib
Description: Vz/F was the apparent volume of distribution after oral dose. It was determined as dose/(AUCinf × kel), where kel was the terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration time curve. The geometric coefficient of variation was reported as percentage.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
Number analyzed (Participants) | 21 | 20 | 4
liter | 11130 (25) | 10650 (24) | 12870 (19)

7. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Bosutinib
Description: t½ was the terminal elimination plasma half-life. It was determined as Loge(2)/kel, where kel was the terminal elimination phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: Predose (0 hour) and at 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 60, 72, 96, and 144 hours post bosutinib dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
Number analyzed (Participants) | 21 | 20 | 4
hour | 47.22 (11.753) | 46.01 (13.434) | 43.28 (7.6939)

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities (Without Regard to Baseline Abnormality)
Description: Laboratory tests included hematology tests, chemistry tests, and urinalysis tests. Laboratory parameters with at least 1 occurrence meeting the pre-defined criteria are reported for this outcome measure.
Time Frame: On Days 4, 5, 7 of Periods 1 and 2 for all participants, on Period 3 Days 4, 5, 7 for participants who were assigned to treatment sequences A=>B=>C and B=>A=>C, and at early termination/discontinuation (if applicable)
Population: All participants randomly assigned to study intervention and who take at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
Number analyzed (Participants) | 30 | 31 | 12
Participants
  Monocytes/Leukocytes (%) >1.2*upper normal limit (ULN) | 7 | 8 | 3
  Aspartate Aminotransferase (U/L) > 3.0*ULN | 1 | 0 | 0
  Creatine Kinase (U/L) >2.0* ULN | 1 | 0 | 0
  Urobilinogen (EU/dL) ≥1 | 1 | 1 | 0
  Coronavirus 19 Molecular (Scalar) >0 | 1 | 2 | 1
  Specific Gravity (scalar) <1.003 | 0 | 2 | 0
  Specific Gravity (scalar) >1.030 | 1 | 0 | 0
  URINE Hemoglobin ≥1 | 4 | 4 | 0
  URINE Bilirubin ≥1 | 0 | 1 | 0

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs are those with initial onset or that worsen in severity after the first dose of the study medication. All AEs in the table below were TEAEs. An SAE is any untoward medical occurrence at any dose that: results in death; is life threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect; or that is considered to be an important medical event. Severe AEs were defined as AEs that interfered significantly with participant's usual function. Both SAEs and severe AEs were according to the investigator's assessment.
Time Frame: Post first dose on Period 1 Day 1 up to 28 days post the last dose of study intervention (up to a maximum of 75 days)
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
Number analyzed (Participants) | 30 | 31 | 12
Participants
  Particiapnts with TEAEs | 13 | 20 | 5
  Particiapnts with SAEs | 0 | 0 | 0
  Particiapnts with severe AEs | 0 | 0 | 0
  Participants discontinued from study due to adverse events | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Post first dose on Period 1 Day 1 up to 28 days post the last dose of study intervention (up to a maximum of 75 days)
Description: Same event may appear as adverse event (AE) and serious AE, what is presented as distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who were randomized and received at least 1 confirmed dose of investigational product.
Arm/Group | Treatment A: Bosutinib 1*100 mg Capsule Fed | Treatment B: Bosutinib 4*25 mg Capsule Fed | Treatment C: Bosutinib 1*100 mg Capsule Fasted
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/31 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/12
Other Adverse Events (participants affected / at risk) | 13/30 | 20/31 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A: Bosutinib 1*100 mg Capsule Fed (N=30) | Treatment B: Bosutinib 4*25 mg Capsule Fed (N=31) | Treatment C: Bosutinib 1*100 mg Capsule Fasted (N=12)
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 1
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 1
Feeling cold (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Electric shock (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 6 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT05032690/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT05032690/SAP_001.pdf